CLINICAL TRIAL: NCT02316977
Title: Home Monitoring of Patients With Chronic Diseases - an eRehab Test-retest Study
Acronym: eRehab
Status: Completed | Type: Observational
Sponsor: Eva Ejlersen Wæhrens (Other)
Responsible Party: Sponsor-Investigator, Eva Ejlersen Wæhrens, Senior researcher, PhD, Parker Research Institute
Organization: Parker Research Institute (Other)
Other Study IDs: 133.1
Record Dates: First submitted 2014-12-08; First posted 2014-12-15 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: Reproducibility of Results
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the study is to establish the intrarater-reliability, criterion validity and responsiveness of the ADL-Questionnaire applied on an eHealth platform to be used by patients diagnosed with rheumatoid arthritis.

The study is designed as a repeated test-retest study including 240 patients filling in the ADL-Q, HAQ-DI and PDQ at day 1, 3, 56 and 58. The study provides an eHealth platform (a home-module in the DANBIO database) which makes it possible for the patients to complete their assessments and send information from their own home.

Intrarater reliability will be assessed by calculating the intraclass correlation coefficients (ICCs). Criterion validity will be evaluated based on correlational analysis and responsiveness based on effect sizes, in both cases involving HAQ-DI. PDQ scores will be used to classify participants based on pain phenotype to explore any relationship between pain phenotype and reliability.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RA ≥ 12 months
* DAS28-CRP < 5,1
* Age between 18 and 85 years
* Computer and Internet connection at home

Exclusion Criteria:

* Blood samples (creatinine, haemoglobin) outside the reference limits +/- 5 % at screening
* Blood samples (thrombocytes and leukocytes) outside the reference limit -/+ 15 % at screening
* Blood samples (ALAT) outside the reference limit -/+ 100 % at screening
* Dementia or other linguistic/cognitive/physical deficiency that prevents participation
* Vision impairment that prevents the use of the devices and computer

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients, diagnosed with RA, referred for regular controls in the rheumatology clinic at Copenhagen University Hospital, Bispebjerg and Frederiksberg, will be screened via the database, DANBIO, for in- and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
ADL-Questionnaire: repeated evaluations to adress reliability, validity and responsiveness | Day 1,3,56 and 58
  Intrarater reliability: day 1-3 and 56-58. Criterion validity: day 1 Responsiveness: day 1-56

SECONDARY OUTCOMES:
Standford Health Assessment Questionnaire Disability Index (HAQ-DI) | Day 1 and 56
  Criterion validity: day 1. Responsiveness: day 1-56
PainDetect Questionnaire (PDQ) | Day 1
  For subgroups analysis

OTHER OUTCOMES:
Disease Activity Score 28 (DAS28) | Day 1,3,56 and 58

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bliddal, DMSci, Study Director — The Parker Research Institute
Locations (1):
- The Parker Research Institute, Department of Rheumatology, Copenhagen University Hospital, Bispebjerg and Frederiksberg, Frederiksberg, Denmark